CLINICAL TRIAL: NCT02030119
Title: A Randomized Trial of Behavioral Economic Interventions to Improve Physical Activities: Framing Incentives
Brief Title: Way to Be Active III (Framing Incentives)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 819149
Record Dates: First submitted 2013-12-20; First posted 2014-01-08 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-09

CONDITIONS: Sedentary Lifestyle
Keywords: Sedentary lifestyle; Pedometers; Obesity; Physical Activity; Financial Incentives; Behavioral Economics
MeSH Terms: conditions — Sedentary Behavior; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Active Comparator): The participant will receive either an email or text message (based on the participant's preference) stating whether the participant achieved their goal for the prior day.
  Interventions: Behavioral: Daily feedback
- Gain Framing (Experimental): Participants will be told that they will earn money for each day they walk at least 7000 steps. Each participant will receive either an email or text message (based on the participant's preference) stating whether or not he/she achieved the goal for the prior day and can collect the earnings. Non-adherent participants will receive messages about how much they would have earned had they met their target step goal.
  Interventions: Behavioral: Financial Incentives; Behavioral: Daily feedback
- Loss Framing (Experimental): The participants will be told that their account has been credited a certain amount of money for the upcoming 30 days. However, for each day they do not meet their goal of at least 7000 steps, they will lose a small portion of that money. The participant will receive either an email or text message (based on the participant's preference) stating whether the participant achieved the goal for the prior day. Non-adherent participants will receive messages about how much the participant would have kept had they met the target step goal.
  Interventions: Behavioral: Financial Incentives; Behavioral: Daily feedback
- Daily Lottery (Experimental): Each participant will be entered into a lottery daily, but participants will only be eligible to collect their winnings if they walked at least 7000 steps the day before. Participants will receive either an email or text message (based on the participant's preference) stating whether or not they won the lottery and if they met their target step goal. If both occur, the participant will be told how much money he or she won. Non-adherent participants will receive messages about how much they would have won had they met the target step goal.
  Interventions: Behavioral: Financial Incentives; Behavioral: Daily feedback

INTERVENTIONS:
Behavioral: Financial Incentives
  Arms: Daily Lottery; Gain Framing; Loss Framing
Behavioral: Daily feedback

SUMMARY:
Employers are increasingly looking for opportunities to motivate sedentary employees to become more physically active. Workplace walking programs have had mixed success and typically show most improvement among participants that are already fairly active at a baseline. The goal of this study is to determine whether a financial incentive program can motivate sedentary employees to increase the number of steps they walk per day to meet a minimum threshold.

The primary outcome measure is the proportion of days a minimum activity of 7000 steps or more is achieved. Outcomes will be assessed each week for 3 months using incentives followed by 3 months of follow-up without incentives. Secondary outcomes will include the average steps walked per day.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18.
2. Participant will need an iPhone or Android smartphone to be able to use the Moves App for tracking steps

Exclusion Criteria:

1. A score of "high" on the International Physical Activity Questionnaire (IPAQ) activity level scale
2. BMI less than 27
3. Pregnant or lactating
4. Participation in another physical activity study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Volpp, MD, PhD, Principal Investigator — University of Pennsylvania; Mitesh Patel, MD, MBA, Study Director — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Patel MS, Asch DA, Rosin R, Small DS, Bellamy SL, Heuer J, Sproat S, Hyson C, Haff N, Lee SM, Wesby L, Hoffer K, Shuttleworth D, Taylor DH, Hilbert V, Zhu J, Yang L, Wang X, Volpp KG. Framing Financial Incentives to Increase Physical Activity Among Overweight and Obese Adults: A Randomized, Controlled Trial. Ann Intern Med. 2016 Mar 15;164(6):385-94. doi: 10.7326/M15-1635. Epub 2016 Feb 16. PMID 26881417

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant randomly assigned to the gain-incentive group was later found to be ineligible due to previous enrollment in another physical activity study. One participant randomly assigned to the lottery-incentive group switched to a phone that was not eligible for use before the study began and therefore did not receive the intervention.
Groups:
- Control: The participant will receive either an email or text message (based on the participant's preference) stating whether the participant achieved their goal for the prior day.
  Daily feedback
- Gain Framing: Participants will be told that they will earn money for each day they walk at least 7000 steps. Each participant will receive either an email or text message (based on the participant's preference) stating whether or not he/she achieved the goal for the prior day and can collect the earnings. Non-adherent participants will receive messages about how much they would have earned had they met their target step goal.
  Financial Incentives
  Daily feedback
- Daily Lottery: Each participant will be entered into a lottery daily, but participants will only be eligible to collect their winnings if they walked at least 7000 steps the day before. Participants will receive either an email or text message (based on the participant's preference) stating whether or not they won the lottery and if they met their target step goal. If both occur, the participant will be told how much money he or she won. Non-adherent participants will receive messages about how much they would have won had they met the target step goal.
  Financial Incentives
  Daily feedback
- Loss Framing: The participants will be told that their account has been credited a certain amount of money for the upcoming 30 days. However, for each day they do not meet their goal of at least 7000 steps, they will lose a small portion of that money. The participant will receive either an email or text message (based on the participant's preference) stating whether the participant achieved the goal for the prior day. Non-adherent participants will receive messages about how much the participant would have kept had they met the target step goal.
  Financial Incentives
  Daily feedback
Period: Overall Study
Arm/Group | Control | Gain Framing | Daily Lottery | Loss Framing
Started | 70 | 70 | 71 | 70
Completed | 67 | 68 | 65 | 67
Not Completed | 3 | 2 | 6 | 3
Not completed — Withdrawal by Subject | 3 | 1 | 5 | 3
Not completed — Ineligible (see Pre-assignment Details) | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Gain Framing | Daily Lottery | Loss Framing | Total
Number analyzed (Participants) | 70 | 69 | 70 | 70 | 279
Age, Continuous [Mean (Standard Deviation); unit: years of age] | 39.4 (12.2) | 37.1 (10.9) | 40.3 (11.2) | 41.9 (11.6) | 39.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 55 | 53 | 54 | 217
  Male | 15 | 14 | 17 | 16 | 62
Mean BMI [Mean (Standard Deviation); unit: kg/m^2] | 33.2 (5.3) | 32.6 (4.5) | 33.1 (5.6) | 33.8 (6.8) | 33.2 (5.6)
Median physical activity in the past 7 d, MET-min [Median (Inter-Quartile Range); unit: Metabolic equivalent minutes (MET-min)] — International Physical Activity Questionnaire (IPAQ) was used to calculate the number of metabolic equivalent minutes (MET-min) per participant in the past 7 days. MET-min is the physiologic measure of energy expenditure, with light-intensity activities having an MET<3, moderate-intensity activities having an MET of 3 to 6, and more vigorous-intensity activities with an MET>6. Population: Analysis population (n=279)
  Metabolic equivalent minutes (MET-min) | 2568.8 [1077.0 to 4941.0] | 2812.2 [1408.0 to 4806.0] | 2785.0 [1336.5 to 4965.5] | 2764.5 [933.0 to 4456.0] | 2709.3 [1299.5 to 4896.0]
Race/ethnicity [Count of Participants; unit: Participants]
  White non-Hispanic | 45 | 41 | 44 | 49 | 179
  African American non-Hispanic | 16 | 16 | 16 | 13 | 61
  Other non-Hispanic | 6 | 10 | 7 | 6 | 29
  Hispanic | 3 | 2 | 3 | 2 | 10
Education [Count of Participants; unit: Participants]
  Less than college | 1 | 2 | 2 | 2 | 7
  Some college | 15 | 15 | 13 | 12 | 55
  College graduate | 54 | 52 | 55 | 56 | 217
Marital status [Count of Participants; unit: Participants]
  Single | 27 | 26 | 27 | 25 | 105
  Married | 31 | 31 | 32 | 36 | 130
  Other | 12 | 12 | 11 | 9 | 44
Annual household income [Count of Participants; unit: Participants]
  <$50,000 | 21 | 24 | 24 | 15 | 84
  $50,000-$100,000 | 25 | 32 | 22 | 29 | 108
  >$100,000 | 20 | 12 | 20 | 18 | 70
Number of Participants with iPhone smartphone [Count of Participants; unit: Participants] | 46 | 43 | 45 | 49 | 183

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Days Each Individual Walks 7000 Steps Per Day or More
Description: The primary outcome measure is the mean proportion of participant-days a minimum activity of 7000 steps or more is achieved. Outcomes will be assessed each week for 3 months using incentives followed by 3 months of follow-up without incentives.
Time Frame: Throughout the 6 month study
Measure: Mean (95% Confidence Interval); unit: Proportion of participant-days
Arm/Group | Control | Gain Framing | Daily Lottery | Loss Framing
Number analyzed (Participants) | 70 | 69 | 70 | 70
Proportion of participant-days
  Intervention | 0.30 [0.22 to 0.37] | 0.35 [0.28 to 0.42] | 0.36 [0.29 to 0.43] | 0.45 [0.38 to 0.52]
  Follow-up | 0.24 [0.18 to 0.31] | 0.25 [0.19 to 0.31] | 0.23 [0.17 to 0.30] | 0.30 [0.24 to 0.37]

2. Secondary Outcome: Average Number of Steps Per Day
Description: Secondary outcomes include average number of steps each individual takes per day throughout the 13-week intervention and additional 13-week follow-up periods.
Time Frame: Throughout the 6 month study
Measure: Mean (95% Confidence Interval); unit: Steps per day
Arm/Group | Control | Gain Framing | Daily Lottery | Loss Framing
Number analyzed (Participants) | 70 | 69 | 70 | 70
Steps per day
  Intervention | 5031 [4406 to 5656] | 5406 [4799 to 6013] | 5251 [4625 to 5876] | 5880 [5265 to 6497]
  Follow-up | 4539 [3916 to 5162] | 4692 [4084 to 5301] | 4529 [3901 to 5158] | 5065 [4466 to 5664]

ADVERSE EVENTS:
Arm/Group | Control | Gain Framing | Daily Lottery | Loss Framing
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/69 | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/69 | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/69 | 0/70 | 0/70

LIMITATIONS AND CAVEATS:
Subjects were from single Philadelphia employer; ppts were required to have a smartphone, and their physical activity was not tracked when they did not have smartphone on them; we did not collect baseline data for step counts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No